CLINICAL TRIAL: NCT00987233
Title: A Study Comparing the Bioequivalence of Triamcinolone Acetonide Aqueous Nasal Spray (Apotex, Inc.) to That of Nasacort® AQ Nasal Spray (Sanofi-Aventis Pharmaceutical Products, Inc.) In the Treatment of Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Apotex Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRIA-NASO-05RB02-CE
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2009-09-30 (Estimated); Status verified 2009-09

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- triamcinolone acetonide aqueous nasal spray (Experimental)
  Interventions: Drug: triamcinolone acetonide aqueous nasal spray (Apotex Inc.)
- Nasacort® AQ Nasal Spray (Active Comparator)
  Interventions: Drug: triamcinolone acetonide aqueous nasal spray (Nasacort® AQ)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: triamcinolone acetonide aqueous nasal spray (Apotex Inc.) — It is to be self-administered; the dosing regimen will be 2 sprays (actuations) into each nostril, once daily. This is the dosing regimen during placebo lead-in and randomized treatment phases. Each actuation of active treatment is equivalent to 55 ug of triamcinolone acetonide, for a total daily dose of 220ug triamcinolone acetonide per day.
  Arms: triamcinolone acetonide aqueous nasal spray
Drug: triamcinolone acetonide aqueous nasal spray (Nasacort® AQ) — It is to be self-administered; the dosing regimen will be 2 sprays (actuations) into each nostril, once daily. This is the dosing regimen during placebo lead-in and randomized treatment phases. Each actuation of active treatment is equivalent to 55 ug of triamcinolone acetonide, for a total daily dose of 220ug triamcinolone acetonide per day.
  Arms: Nasacort® AQ Nasal Spray
Drug: Placebo — It is to be self-administered; the dosing regimen will be 2 sprays (actuations) into each nostril, once daily. This is the dosing regimen during placebo lead-in and randomized treatment phases. Each actuation of active treatment is equivalent to 55 ug of triamcinolone acetonide, for a total daily dose of 220ug triamcinolone acetonide per day.
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled parallel-group study, comparing the bioequivalence of triamcinolone acetonide aqueous nasal spray (Apotex, Inc.) to that of Nasacort® AQ nasal spray (Sanofi-Aventis Pharmaceutical Products, Inc.) in the treatment of seasonal allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Understands the requirements of the study and provides written informed consent;
* Is a male or female between 18 and 65 years of age;
* At least a 2-year history of seasonal allergic rhinitis;
* The presence of IgE-mediated hypersensitivity to local pollen confirmed by a positive response to either skin prick or intradermal testing within the past 12 months. A positive response is defined as a wheal diameter of at least 3 mm larger than the control for the skin prick test or at least 7 mm larger than the control for the intradermal test;
* In order to enter the placebo lead-in period, the subject must have a score of at least 6 on a 24-hour reflective TNSS completed during Visit 2;
* Is in general good health as determined by screening evaluations and the judgment of the Investigator;
* If female of childbearing potential, is not pregnant (confirmed by negative urine pregnancy test), non-lactating, and will use reliable birth control measures throughout the study. Female of child bearing potential is defined as a female who has experienced menarche, and who has not undergone successful surgical sterilization: hysterectomy, bilateral oophorectomy or ovariectomy, bilateral tubal ligation or salpingectomy; or is not postmenopausal for at least 1 year.;
* If receiving immunotherapy, must be on a stable maintenance regimen for at least 30 days before Visit 1, and should maintain the same dose throughout the study (Low dose antibiotic therapy given prophylactically and started prior to Day -7 is acceptable.);
* Has not used systemic steroids or topical steroids (inhaled, intranasal, or intraocular) within 30 days before Visit 2; Is capable of tolerating intranasal application of the study drug; and
* Is willing and able to comply with the requirements of the protocol and intends to complete the study.

Exclusion Criteria:

* Evidence of any unstable or clinically significant, hematopoietic, malignant, cardiovascular, hepatic, renal, neurologic, psychiatric, or autoimmune disorder/condition/disease that in the opinion of the Investigator could place the subject at increased risk of complications, interfere with study participation, or confound any of the study objectives;
* Presence or history of ocular herpes simplex, cataracts, or glaucoma;
* Inability to avoid exposure to chickenpox or measles;
* Respiratory tract infection within two weeks prior to screening;
* Infection requiring oral antibiotic treatment two weeks prior to screening;
* Significant pulmonary disease and/or active asthma requiring daily medication;
* Signs or symptoms of nasal polyps, deviated septum, or any other condition, which in the opinion of the Investigator, may result in erroneous study data; Known intolerance (hypersensitivity or serious adverse reaction) to corticosteroids;
* History within the last 5 years or current evidence of alcohol or drug abuse;
* Current use of therapies or medications (e.g., tricyclic antidepressants and others. See Section 8.1, Prohibited Medications) that would affect assessment of the effectiveness of the study drugs;
* Unable to withhold any prohibited medication (see Section 8.1, Prohibited Medications);
* Use of any of the following prior to the start of the single-blind placebo lead-in visit (Visit 2) within the time periods specified:

Time prior to Visit 2

* Intranasal or systemic corticosteroids 30 days
* Ocular corticosteroids 30 days
* Intranasal cromolyn 14 days
* Leukotriene inhibitors 14 days
* Loratadine10 days
* Intranasal or systemic antihistamines (including sleep and diet aids and cold preparations) 3 days
* Has received any investigational drug or participated in an investigational research study within 30 days of entering this study;
* Documented evidence of acute or significant chronic sinusitis, as determined by the investigator;
* Rhinitis medicamentosa;
* Planned travel outside the study area for a substantial portion of the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
To demonstrate similar efficacy (bioequivalence) of the generic triamcinolone acetonide aqueous nasal spray (Apotex, Inc.) with that of the marketed reference drug, Nasacort® AQ Nasal Spray in the treatment of seasonal allergic rhinitis.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinsys Clinical Research, Inc., Bedminster, New Jersey, United States